CLINICAL TRIAL: NCT05675631
Title: Effects of Suspension Training Versus a Traditional One in the Elderly Population: a Randomized Clinical Trial
Brief Title: Effects of Suspension Training in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, David Hernández-Guillén, Assistant professor, PT, PhD, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: OA_SUSTRAIN
Record Dates: First submitted 2022-12-29; First posted 2023-01-09 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Old Age; Atrophy
Keywords: Suspension; Older adult; Balance; Strength; Prevention
MeSH Terms: conditions — Atrophy | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): This group will perform training using suspension elements.
  Interventions: Other: Suspension training
- Control Group (Active Comparator): This group will perform training using weights and elastic bands.
  Interventions: Other: Strength training

INTERVENTIONS:
Other: Suspension training — This group will perform training using suspension devices.
  Arms: Experimental Group
Other: Strength training — This group will perform training using weights and elastic bands.
  Arms: Control Group

SUMMARY:
Traditionally, tools that use unstable surfaces have been used to increase the difficulty of exercises by stimulating the recruitment of a greater number of motor units. A new method is suspension training. It uses the weight of the body and the principles of moments of forces to improve the recruitment of motor units. The difficulty that stimulates this recruitment depends on the amount of instability caused by the suspension apparatus and the position of the body.

So this type of training in the elderly can be very interesting due to the ease of adaptation, since it can be used as a facilitating method or to increase the difficulty.

It seems that suspension training can have positive effects that will have a direct impact on the quality of life of the elderly, due to improvements in different aspects such as gaining strength and improving balance, consequently reducing the risk of falling. . It is a good alternative to gain strength and improve functional mobility and upper trunk strength in the elderly, to other exercises such as elastic bands, since they produce similar effects.

For all these reasons, the program tries to demonstrate that suspension training can be an effective tool to improve the quality of life and reduce the risk of falls in the elderly.

DETAILED DESCRIPTION:
This research originates from the curiosity of wanting to prove that exercise in the elderly is more than recommended, specifically suspension training.

Traditionally, tools that use unstable surfaces have been used to increase the difficulty of exercises by stimulating the recruitment of a greater number of motor units. A new method is suspension training. It uses the weight of the body and the principles of moments of forces to improve the recruitment of motor units. The difficulty that stimulates this recruitment depends on the amount of instability caused by the suspension apparatus and the position of the body.

So this type of training in the elderly can be very interesting due to the ease of adaptation, since it can be used as a facilitating method or to increase the difficulty.

Additionally, an unstable resistance training situation stresses/taxes the neuromuscular system and can promote a greater gain in strength and increase the cross-sectional area. It can also increase motor unit recruitment and improve neuromuscular coordination without an increase in mechanical load when performing push-ups under unstable conditions. Because TRX exercises involve normal resistance, they can potentially improve strength by facilitating the use of large and fast-twitch muscle units, increasing muscle coordination and stimulating the musculoskeletal system, and increasing the number of muscle fibers. Suspension work increases the activation of most muscle groups involved in suspension training (push-ups, inverted row, prone bridge and hamstring curl) compared to traditional training.

Likewise, for the upper extremity it improves significantly as well as training with elastic bands. Improves the handgrip. Due to the constant use of suspension elements. For the lower extremity, a very high activation of the biecps femoris and semitendinosus (<90% MVIC), hamstrings, gluteus maximus, gluteus medius and adductor lagus have been observed. In relation to balance, it has been observed that suspension training has more notable positive effects on it than in traditional training due to the constant adaptation and participation of the CORE in the different exercises. On the other hand, regarding the fear of falls, it has been observed that, in medium and high intensity programs, this fear decreases as the participants feel more confident. In this type of study, positive effects have also been shown on sleep quality through the PSQI, positive effects on stride after high intensity and positive changes in body composition: higher percentage of water at the cellular level, with which better value of PhA and better cellular health. Finally, another possible advantage is the ease of installation of the material and its affordable price, since traditional training often requires more expensive machines and tools.

It seems then that suspension training can have positive effects that will have a direct impact on the quality of life of the elderly, due to improvements in different aspects such as gaining strength and improving balance, consequently reducing the risk of suffering a drop. It is a good alternative to gain strength and improve functional mobility and upper trunk strength in the elderly, to other exercises such as elastic bands, since they produce similar effects.

For all these reasons, the program tries to demonstrate that suspension training can be an effective tool to improve the quality of life and reduce the risk of falls in the elderly.

ELIGIBILITY:
Inclusion Criteria:

* Older adults between 60 and 85 years

Exclusion Criteria:

* Not wanting to sign the informed consent.
* Present pathology of the central nervous system that negatively affects balance, strength or compression; or cardiac pathologies in which strength exercise is contraindicated.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Hand Grip Test | Baseline (0 week)
  Grip strength is usually measured using a hand-held dynamometer. The patient squeezes the dynamometer with all of their strength, typically three times with each hand. An average score is then calculated using the measurements from both hands.
Hand Grip Test | Post-treatment (7 week)
  Grip strength is usually measured using a hand-held dynamometer. The patient squeezes the dynamometer with all of their strength, typically three times with each hand. An average score is then calculated using the measurements from both hands.

SECONDARY OUTCOMES:
5 Times Sit-to-Stand Test | Baseline (0 week), post-treatment (7 week)
  Assesses functional lower extremity strength, transitional movements, balance, and fall risk. Equipment: Stopwatch; standard height chair with straight back (16 inches high); Therapist Instructions: Have the patient sit with their back against the back of the chair. he test provides a method to quantify functional lower extremity strength and/or identify movement strategies a patient uses to complete transitional movements.The time it takes to do it is timed.
One leg balance | Baseline (0 week), post-treatment (7 week)
  Monopodal balance, count the time you can stand on one leg. The longer the time, the better the equilibrium state.
Functional Reach | Baseline (0 week), post-treatment (7 week)
  Functional range that consists of measuring how much the participant can move or lean forward without losing stability. The greater the distance, the greater the stability.
Test Get-Up and Go | Baseline (0 week), post-treatment (7 week)
  Dynamic or functional balance in which the time it takes to get up, travel a distance of 3m round trip and return to sit down is timed. The less time, the better functional status.
Walking speed test | Baseline (0 week), post-treatment (7 week)
  The speed of the step is calculated by means of the chrono of what it takes to cover a distance of 4 meters. The higher the walking speed, the better the prognosis.
Quality of live (EQ-5D) | Baseline (0 week), post-treatment (7 week)
  The EQ-5D-5L is a self-assessed, health related, quality of life questionnaire. The scale measures quality of life on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The lower the score on the questions, the better the status will be. On the analog scale, the higher the score, the better the state of health.
Falls Efficacy Scale International | Baseline (0 week), post-treatment (7 week)
  The Falls Efficacy Scale-International (FES-I) is a short, easy to administer tool that measures the level of concern about falling during 16 social and physical activities inside and outside the home whether or not the person actually does the activity.

CONTACTS AND LOCATIONS:
Overall Officials: David Hernández-Guillén, PT, PhD, Principal Investigator — University of Valencia
Locations (1):
- University of Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No